CLINICAL TRIAL: NCT05094375
Title: Vaginal Misoprostol 600 mcg and 800 mcg In Medical Treatment of First Trimester Missed Miscarriage: A Randomized Controlled Trial.
Brief Title: Vaginal Misoprostol In Medical Treatment of First Trimester Missed Miscarriage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: hany farouk (Other)
Responsible Party: Sponsor-Investigator, hany farouk, Clinical Professor, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aswu/354/10/19
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Miscarriage
Keywords: miscarriage; vaginal; misoprostol
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Intervention Model Description: a double-blinded randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a double-blinded randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Misoprostol 600 mcg (Experimental): All patients will receive three doses of vaginal misoprostol every four hours. The first dose of misoprostol 600 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  * Two doses of misoprostol 600 mcg each (3 tablets of 200 mcg per dose).
  * Paracetamol, eight hourlies, will be provided as analgesic or antipyretic.
  * A specimen bottle to collect the POC if passed out.
  * Two pairs of disposable gloves.
  * Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Interventions: Drug: Vaginal Misoprostol 600 mcg
- Vaginal Misoprostol 800 mcg (Active Comparator): All patients will receive three doses of vaginal misoprostol every four hours. The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  * Two doses of misoprostol 800 mcg each (four tablets of 200 mcg per dose).
  * Paracetamol, eight hourlies, will be provided as analgesic or antipyretic.
  * A specimen bottle to collect the POC if passed out.
  * Two pairs of disposable gloves.
  * Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Interventions: Drug: Vaginal Misoprostol 800 mcg

INTERVENTIONS:
Drug: Vaginal Misoprostol 600 mcg — All patients will receive three doses of vaginal misoprostol every four hours. The first dose of misoprostol 600 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  * Two doses of misoprostol 600 mcg each (3 tablets of 200 mcg per dose).
  * Paracetamol, eight hourlies, will be provided as analgesic or antipyretic.
  * A specimen bottle to collect the POC if passed out.
  * Two pairs of disposable gloves.
  * Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Other Names: experimental
  Arms: Vaginal Misoprostol 600 mcg
Drug: Vaginal Misoprostol 800 mcg — All patients will receive three doses of vaginal misoprostol every four hours. The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of second dose will be given upon sending home.
  * Two doses of misoprostol 800 mcg each (four tablets of 200 mcg per dose).
  * Paracetamol, eight hourlies, will be provided as analgesic or antipyretic.
  * A specimen bottle to collect the POC if passed out.
  * Two pairs of disposable gloves.
  * Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Other Names: Active Comparator
  Arms: Vaginal Misoprostol 800 mcg

SUMMARY:
Efficacy of vaginal misoprostol 600 Mg versus 800 Mg in termination of the first trimester missed abortion were assist

DETAILED DESCRIPTION:
In women with first trimetric-missed miscarriage, vaginal misoprostol in the achievement of successful miscarriage so our aim was to compare the effectiveness of vaginal misoprostol 600 Mg versus 800 Mg for medical treatment of the first trimester missed miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* All women above 18 years of age
* Less than 12 weeks of gestation.
* Pregnancy is confirmed by pregnancy test or ultrasound scan.
* missed abortion
* Normal general and gynecological examination.

Exclusion Criteria:

* Hemodynamically unstable.
* Suspected sepsis with temperature 38 °C.
* Concurrent medical illness e.g. hematological, cardiovascular, thromboembolism,
* respiratory , recent liver disease, or pruritus of pregnancy.
* Presence of intrauterine contraceptive device (IUCD).
* Suspect or proven ectopic pregnancy.
* Failed medical or surgical evacuation before the presentation.
* Known allergy to misoprostol.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with missed abortion
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Completeness of abortion | 7 days
  expulsion of Products of conception by visual inspection

SECONDARY OUTCOMES:
Successful medical abortion | 14 days
  cervical os is closed with endometrial thickness of less than 15 mm
Bleeding pattern following treatment | 7 days
  This will be assessed by hemoglobin(g/dl) and haematocrit level after the treatment , if the patients required blood transfusion and number of units transfused and number of days of bleeding
Pain resulting from the procedure | 7 days
  this will be assessed by the doses of paracetamol given in mg
Additional uterotonic used | 14 days
  additional misoprostol doses in mcg

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No